CLINICAL TRIAL: NCT04133519
Title: The Efficacy and Safety of IBS Digital Behavioral Treatment Study
Brief Title: Efficacy and Safety of IBS Digital Behavioral Treatment
Acronym: EASITx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: metaMe Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM001
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS - Irritable Bowel Syndrome; IBS; Irritable Bowel
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Neuromuscular Blockade

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Comparator-Controlled, Parallel-Group Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Arm 1 is an active behavioral treatment for IBS (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD).
  Interventions: Device: Arm 1 - Active behavioral Treatment Arm (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD)
- Arm 2 (Active Comparator): Arm 2 is a behavioral treatment (MR-1; Muscle Relaxation, Software as a Medical Device - SaMD)
  Interventions: Device: Arm 2 - Active Comparator behavioral treatment arm (MR-1; Muscle Relaxation, Software as a Medical Device - SaMD)

INTERVENTIONS:
Device: Arm 1 - Active behavioral Treatment Arm (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD) — The active treatment consists of 7 unique video/audio recordings administered via a mobile application every other week for 12 weeks (SaMD). Since subjects in both the active and comparator treatment arms receive a behavioral treatment, the subjects are blinded to active treatment.
  Arms: Arm 1
Device: Arm 2 - Active Comparator behavioral treatment arm (MR-1; Muscle Relaxation, Software as a Medical Device - SaMD) — The comparator treatment consists of an identical treatment platform, scheduling platform, and reminder platform as the Active Treatment Arm, but in place of Gut-Directed Hypnotherapy there is a comparator relaxation treatment administered on an identical schedule: 7 unique video/audio recordings administered via a mobile application every other week for 12 weeks.
  Arms: Arm 2

SUMMARY:
A Randomized, Double-Blind, Comparator-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Two Self-administered behavioral treatments for Adult Subjects with Symptomatic Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
EASITx is a pivotal study comparing two self-administered behavioral treatments for irritable bowel syndrome (IBS). The active treatment in EASITx is classified as Software as a Medical Device (SaaMD).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-70
* Confirmation of the IBS and IBS subtype diagnosis by a study site physician using Rome IV diagnostic criteria
* Possess an iPhone Operating System (iOS) Apple or Android smartphone or iOS tablet (iPad) released in 2015 or later
* Agreement to input information about their abdominal pain and bowel movements on a daily basis into Curebase software
* Agreement to have their anonymized data stored in the cloud for up to 2 years after the conclusion of the study, and to have the data used for research purposes.
* Agreement to maintain stable dosage of IBS medications during the course of treatment and not to add new IBS medication or stop current IBS medications unless directed to do so by the participants treating physician. Changes in treatment will be captured using a concomitant medication assessment.
* Average "Worst Daily Pain Severity" of >3 on a 11-point numeric rating scale (NRS) over the full 28-day pre-treatment symptom tracking period
* Consistent submission of Pain Severity scores via the Curebase app (data submitted on 80% or more of days in the symptom tracking window)

Exclusion Criteria:

* Evidence of current structural intestinal abnormalities that better explain the participant's IBS symptoms (e.g., celiac disease, inflammatory bowel disease - Crohn's Disease and ulcerative colitis, prior abdominal surgeries such as weight loss surgery or bowel resection)
* Medication use, other illnesses or conditions that can explain their gastrointestinal symptoms e.g.,regular narcotic use or dependency, Over The Counter (OTC) stimulant laxative dependence (i.e, progressively larger doses of Senna or Bisacodyl containing compounds are needed to produce a bowel movement), history of radiation to the abdomen.
* Diagnosed and/or treated for a malignancy within the past 5 years (other than localized basal or squamous cell carcinomas of the skin)
* Current psychotherapy, hypnotherapy, or cognitive behavioral therapy (CBT) for IBS
* Inability to commit to completing all treatment sessions
* Have an unstable extraintestinal condition whose immediate or foreseeable treatment needs would realistically interfere with study demands, e.g., ability to participate in online treatment sessions or follow daily diary.
* Active psychiatric disorder (e.g., post-traumatic stress disorder, depression associated with high risk of suicidal behavior, psychotic or delusional disorders, dissociative disorders, or gross cognitive impairment)
* Subjects that report a current gastrointestinal infection or an infection within the 4 weeks prior to the evaluation that would otherwise obscure IBS symptoms. In cases of gastrointestinal infection baseline evaluation will be delayed a minimum of 4 weeks until after complete recovery.
* Current or recent use of a gut-targeted antibiotic such as Neomycin or Rifaximin during the 12 weeks prior to baseline assessment. In the case of treatment with rifaximin or neomycin, eligibility will be suspended for 12 weeks from the initial date of use.
* Any condition that an investigator feels may interfere with the conduct of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Pun, DO, Principal Investigator — Elevated Health
Locations (1):
- Curebase, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Serag HB. Impact of irritable bowel syndrome: prevalence and effect on health-related quality of life. Rev Gastroenterol Disord. 2003;3 Suppl 2:S3-11. PMID 12775997
- [Background] Ford AC, Bercik P, Morgan DG, Bolino C, Pintos-Sanchez MI, Moayyedi P. Validation of the Rome III criteria for the diagnosis of irritable bowel syndrome in secondary care. Gastroenterology. 2013 Dec;145(6):1262-70.e1. doi: 10.1053/j.gastro.2013.08.048. Epub 2013 Aug 28. PMID 23994201
- [Background] Leong SA, Barghout V, Birnbaum HG, Thibeault CE, Ben-Hamadi R, Frech F, Ofman JJ. The economic consequences of irritable bowel syndrome: a US employer perspective. Arch Intern Med. 2003 Apr 28;163(8):929-35. doi: 10.1001/archinte.163.8.929. PMID 12719202
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Mayer EA, Tillisch K. The brain-gut axis in abdominal pain syndromes. Annu Rev Med. 2011;62:381-96. doi: 10.1146/annurev-med-012309-103958. PMID 21090962
- [Background] Lackner JM. The role of psychosocial factors in functional gastrointestinal disorders. Quigley, Hongo, Fukuda (eds): Functional and GI Motility Disorders. 2014(33):104-16.
- [Background] Lacy BE, Patel H, Guerin A, Dea K, Scopel JL, Alaghband R, Wu EQ, Mody R. Variation in Care for Patients with Irritable Bowel Syndrome in the United States. PLoS One. 2016 Apr 26;11(4):e0154258. doi: 10.1371/journal.pone.0154258. eCollection 2016. PMID 27116612
- [Background] Blanchard EB, Greene B, Scharff L, Schwarz-McMorris SP. Relaxation training as a treatment for irritable bowel syndrome. Biofeedback Self Regul. 1993 Sep;18(3):125-32. doi: 10.1007/BF00999789. PMID 8218507
- [Background] Palsson OS. Hypnosis Treatment of Gastrointestinal Disorders: A Comprehensive Review of the Empirical Evidence. Am J Clin Hypn. 2015 Oct;58(2):134-58. doi: 10.1080/00029157.2015.1039114. PMID 26264539
- [Background] Lackner JM, Jaccard J, Keefer L, Brenner DM, Firth RS, Gudleski GD, Hamilton FA, Katz LA, Krasner SS, Ma CX, Radziwon CD, Sitrin MD. Improvement in Gastrointestinal Symptoms After Cognitive Behavior Therapy for Refractory Irritable Bowel Syndrome. Gastroenterology. 2018 Jul;155(1):47-57. doi: 10.1053/j.gastro.2018.03.063. Epub 2018 Apr 25. PMID 29702118
- [Background] Flik CE, Laan W, Zuithoff NPA, van Rood YR, Smout AJPM, Weusten BLAM, Whorwell PJ, de Wit NJ. Efficacy of individual and group hypnotherapy in irritable bowel syndrome (IMAGINE): a multicentre randomised controlled trial. Lancet Gastroenterol Hepatol. 2019 Jan;4(1):20-31. doi: 10.1016/S2468-1253(18)30310-8. Epub 2018 Nov 23. PMID 30473202
- [Background] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Background] Yeh VM, Schnur JB, Montgomery GH. Disseminating hypnosis to health care settings: Applying the RE-AIM framework. Psychol Conscious (Wash D C). 2014 Jun;1(2):213-228. doi: 10.1037/cns0000012. PMID 25267941
- [Background] Gonsalkorale WM, Miller V, Afzal A, Whorwell PJ. Long term benefits of hypnotherapy for irritable bowel syndrome. Gut. 2003 Nov;52(11):1623-9. doi: 10.1136/gut.52.11.1623. PMID 14570733
- [Background] Lowen MB, Mayer EA, Sjoberg M, Tillisch K, Naliboff B, Labus J, Lundberg P, Strom M, Engstrom M, Walter SA. Effect of hypnotherapy and educational intervention on brain response to visceral stimulus in the irritable bowel syndrome. Aliment Pharmacol Ther. 2013 Jun;37(12):1184-97. doi: 10.1111/apt.12319. Epub 2013 Apr 25. PMID 23617618
- [Background] Powell RA, Gee TL. The effects of hypnosis on dissociative identity disorder: a reexamination of the evidence. Can J Psychiatry. 1999 Nov;44(9):914-6. doi: 10.1177/070674379904400908. PMID 10584162
- [Background] Meyerson J, Konichezy A. Out-of-illness experience: hypnotically induced dissociation as a therapeutic resource in treating people with obstinate mental disorders. Am J Psychother. 2009;63(2):133-46. doi: 10.1176/appi.psychotherapy.2009.63.2.133. PMID 19711767
- [Background] Hauser W, Hagl M, Schmierer A, Hansen E. The Efficacy, Safety and Applications of Medical Hypnosis. Dtsch Arztebl Int. 2016 Apr 29;113(17):289-96. doi: 10.3238/arztebl.2016.0289. PMID 27173407
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Bang H, Flaherty SP, Kolahi J, Park J. Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol. Clin Res and Reg Affairs, 2010;27(2):42-51
- [Background] Williamson A. What is hypnosis and how might it work? Palliat Care. 2019 Jan 31;12:1178224219826581. doi: 10.1177/1178224219826581. eCollection 2019. No abstract available. PMID 30728719
- [Background] Palsson OS. Standardized hypnosis treatment for irritable bowel syndrome: the North Carolina protocol. Int J Clin Exp Hypn. 2006 Jan;54(1):51-64. doi: 10.1080/00207140500322933. PMID 16316883
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Palsson OS, Baggish JS, Turner MJ, Whitehead WE. IBS patients show frequent fluctuations between loose/watery and hard/lumpy stools: implications for treatment. Am J Gastroenterol. 2012 Feb;107(2):286-95. doi: 10.1038/ajg.2011.358. Epub 2011 Nov 8. PMID 22068664
- [Derived] Berry SK, Berry R, Recker D, Botbyl J, Pun L, Chey WD. A Randomized Parallel-group Study of Digital Gut-directed Hypnotherapy vs Muscle Relaxation for Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2023 Nov;21(12):3152-3159.e2. doi: 10.1016/j.cgh.2023.06.015. Epub 2023 Jun 28. PMID 37391055

RESULTS

PARTICIPANT FLOW:
Groups:
- Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD: Arm 1 is an active behavioral treatment for Irritable Bowel Syndrome (IBS) (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD).
  Arm 1 - Active behavioral Treatment Arm (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD): The active treatment consists of 7 unique video/audio recordings administered via a mobile application every other week for 12 weeks (SaMD). Since subjects in both the active and comparator treatment arms receive a behavioral treatment, the subjects are blinded to active treatment.
- MR-1; Muscle Relaxation, Software as a Medical Device - SaMD: Arm 2 is a behavioral treatment (MR-1; Muscle Relaxation, Software as a Medical Device - SaMD)
  Arm 2 - Active Comparator behavioral treatment arm (MR-1; Muscle Relaxation, Software as a Medical Device - SaMD): The comparator treatment consists of an identical treatment platform, scheduling platform, and reminder platform as the Active Treatment Arm, but in place of Gut-Directed Hypnotherapy there is a comparator relaxation treatment administered on an identical schedule: 7 unique video/audio recordings administered via a mobile application every other week for 12 weeks.
Period: Overall Study
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Started | 188 | 190
Completed | 182 | 184
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Never started treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: 16 participants in the safety analysis population were excluded from the efficacy analysis population (baseline participants); 8 were excluded for being under age 22 (4 in each treatment group), and 7 participants (4 in the MR group and 3 in the GDH group) did not meet eligibility criteria or experienced technical issues with the Curebase software that prevented study execution. Additionally, 2 participants (1 in each group) were excluded because they did not begin a treatment session.
Groups:
- Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD: Arm 1 is an active behavioral treatment for IBS (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD).
  Arm 1 - Active behavioral Treatment Arm (Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD): The active treatment consists of 7 unique video/audio recordings administered via a mobile application every other week for 12 weeks (SaMD). Since subjects in both the active and comparator treatment arms receive a behavioral treatment, the subjects are blinded to active treatment.
- Total: Total of all reporting groups
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD | Total
Number analyzed (Participants) | 181 | 181 | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.1) | 42.6 (12.2) | 42.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 145 | 289
  Male | 37 | 36 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 14 | 16 | 30
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 52 | 59 | 111
  White | 101 | 95 | 196
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 181 | 181 | 362
Baseline abdominal pain intensity [Mean (Standard Deviation); unit: units on a scale] — The Instrument is a 0-10 numeric rating scale (NRS, 0= no pain, 10= worst pain). The subject is asked daily to record their "worst abdominal pain over the past 24-hours". The daily abdominal pain intensity is the average daily pain intensity over the 4 weeks of phase 1 (weeks -4 through -1) before the start of treatment.
  units on a scale | 5.5 (1.75) | 5.4 (1.60) | 5.4 (1.68)
Baseline abdominal pain frequency [Mean (Standard Deviation); unit: days per week] — Baseline average abdominal pain frequency is defined as the average number of days per week during the 4-week pre-treatment assessment period (Week -4 to -1) in which the subjects recorded a 1 or greater on the daily pain intensity measurement. Only days during which an assessment is recorded was included in the calculation of average baseline abdominal pain frequency. Days where severity was >0 were considered a day with pain and were recorded as positive. Days with a score of 0 were days without pain. Mean represents the mean number of days per week with abdominal pain.
  days per week | 6.8 (0.47) | 6.8 (0.42) | 6.8 (0.44)
Baseline IBS-Quality of Life score [Mean (Standard Deviation); unit: units on a scale] — The IBS QOL is a 34 item IBS-specific, validated instrument. The 34 item patient responses are summed for a total score and then transformed to 0-100 scale with higher scores indicating better IBS specific quality of life. The IBS QOL questionnaire was completed by patients once at Week -4 prior to treatment and the baseline score calculated based on these responses.
  units on a scale | 54.7 (20.89) | 51.1 (21.19) | 52.9 (21.08)
IBS with constipation (IBS-C) [Count of Participants; unit: Participants] — The IBS-C subtype designation is based on a diagnosis by a study physician using Rome IV diagnostic criteria
  Participants | 60 | 62 | 122
IBS with diarrhea (IBS-D) [Count of Participants; unit: Participants] — The IBS-D subtype designation is based on a diagnosis by a study physician using Rome IV diagnostic criteria
  Participants | 62 | 60 | 122
IBS with mixed bowel habits (IBS-M) [Count of Participants; unit: Participants] — The IBS-M subtype designation is based on a diagnosis by a study physician using Rome IV diagnostic criteria
  Participants | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Pain Intensity Responder
Description: The primary endpoint of this study is abdominal pain intensity. The Instrument is a 0-10 numeric rating scale (NRS, 0= no pain, 10= worst pain). The subject is asked daily to record their "worst abdominal pain over the past 24-hours".
  An Abdominal Pain Intensity Responder is defined as a subject whose daily abdominal pain intensity averaged over the 4 weeks post-treatment (weeks 13 through 16) is at least 30% reduced compared to the daily abdominal pain intensity averaged over the 4 weeks pre-treatment (weeks -4 through -1).
Time Frame: Baseline score (average of daily score for weeks -4 through -1) was compared to 4-weeks post-treatment (average daily score for weeks 13 through 16)
Population: 16 participants in the safety analysis population were excluded from the efficacy analysis population; 8 were excluded for being under age 22 (4 in each treatment group), and 7 participants (4 in the MR group and 3 in the GDH group) did not meet eligibility criteria or experienced technical issues with the Curebase software that prevented study execution. Additionally, 2 participants (1 in each group) were excluded because they did not begin a treatment session.
Measure: Count of Participants; unit: Participants
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 181 | 181
Participants | 55 | 49
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; P value from Cochran-Mantel-Haenszel testing of H0: OR=1; H1: OR≠1 adjusting for IBS subtype and gender; Test type: Superiority; p = 0.5352, Cochran-Mantel-Haenszel — P value from Cochran-Mantel-Haenszel testing of H0: OR=1; H1: OR≠1 adjusting for IBS subtype and gender; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.73 to 1.84]
Statistical Analysis 2: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The final 4 weeks of the on-treatment period (weeks 9-12) was a pre-specified period for analysis of the primary endpoint measure of abdominal pain due to IBS. An abdominal pain intensity responder was defined as a participant whose daily abdominal pain intensity averaged over the last 4 weeks of phase s (weeks 9 through 12) was at least 30% reduced compared with the daily abdominal pain intensity averaged over the 4 weeks of phase 1; Test type: Superiority; p = 0.0232, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.08 to 2.87] — Odds ratio reflects the odds of the number of GDH responders being greater than the number of MR responders for abdominal pain intensity
Statistical Analysis 3: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; Abdominal pain scores were averaged each week on treatment (1-12) and compared with the average baseline abdominal pain score. Participants that recorded a > 30% decrease in abdominal pain in at least half the weeks on treatment were considered responders. This analysis was specified in FDA Guidance for Industry, "Irritable Bowel Syndrome - Clinical Evaluation of Drugs for Treatment", May 2012. Both the analysis period and the responder threshold (30%) are specified by the FDA Guidance; Test type: Superiority; p = 0.0254, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel Test testing H0: OR=1; H1: OR<>1 adjusting for IBS subtype and gender; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.07 to 2.89] — Odds ratio reflects the odds of GDH being superior to MR; Among all subjects, 64.0% reported Adequate Relief and 67.7% reported overall satisfaction with Regulora

2. Secondary Outcome: Abdominal Pain Intensity
Description: The Instrument is a 0-10 numeric rating scale (NRS, 0= no pain, 10= worst pain). The subject is asked daily to record their "worst abdominal pain over the past 24-hours". Mean change in reported abdominal pain intensity.
Time Frame: as for outcome 1
Population: The analysis population includes all participants with both baseline (weeks -4 to -1 before treatment) and 4-week post treatment period (Weeks 13-16) daily pain scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 168 | 167
units on a scale | -0.995 (1.66) | -1.031 (1.68)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The least square (LS) mean difference between the GDH and MR groups using an analysis of variance (ANOVA) model; Test type: Superiority; p = 0.8115, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.434 to 0.554]

3. Secondary Outcome: Abdominal Pain Frequency
Description: Mean change in reported abdominal pain frequency. The abdominal pain frequency is based on the frequency of abdominal pain measured using a 0-10 numeric rating scale (NRS, 0= no pain, 10= worst pain). The subject is asked daily to record their "worst abdominal pain over the past 24-hours".
  Average abdominal pain frequency is defined as the average number of days per week during the 4-week post-treatment assessment period in which the subjects recorded a 1 or greater on the daily pain measurement. Only days during which an assessment is recorded will be included in the calculation of average abdominal pain frequency. Days where severity was >0 were considered a day with pain and were recorded as positive. Days with a score of 0 were days without pain. Mean represents the mean number of days per week in each time period with abdominal pain. A lower score is a better outcome.
Time Frame: Change from baseline (weeks -4 to -1 before treatment) to 4-week post treatment period (Weeks 13-16)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days/week with abdominal pain
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 171 | 174
days/week with abdominal pain | -0.366 (1.1272) | -0.437 (1.2437)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; Average abdominal pain frequency at Week 13-16 will be statistically compared between GDH and comparator using an ANOVA model adjusted for gender and IBS subtype. The daily pain frequency measurement was derived from the daily pain intensity measurement. Days where severity was >0 were considered a day with pain and were recorded as positive. Days with a score of 0 were days without pain. Mean represents the mean number of days in each time period with abdominal pain; Test type: Superiority; p = 0.7564, ANOVA; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.236 to 0.325]

4. Secondary Outcome: Number of Participants With >=30% Improvement in Normal Bowel Movements (Scored as 3, 4, or 5 on the Bristol Stool Form Scale)
Description: Number of Participants with a ≥ 30% improvement in the proportion of Bristol Stool Form Scale (BSFS) scores that fell within Group 2 (normal stools) compared with baseline (Weeks -4 through -1). The result represents the number of participants with ≥ 30% improvement in the percentage of normal stools The BSFS is a visual aid that allows patients to classify their bowel movements into seven groups ranging from a score of 1 (separate hard lumps) to 7 (watery, no solid pieces). The BSFS scores will be grouped as 1,2 (Group 1), 3,4,5 (Group 2) and 6,7 (Group 3). The mid-range bowel movements 3,4 and 5 (Group 2) define normal stools.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 181 | 181
Participants | 77 | 72
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; A Stool Consistency Responder is defined as a >=30% improvement in the proportion of Bristol Stool Form Scale (BSFS) scores that fall within Group 2 (normal stools); Test type: Superiority; p = 0.4753, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel Test testing H0: OR=1; H1: OR<>1 adjusting for IBS subtype and gender; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.76 to 1.81] — GDH:MR Relative Risk

5. Secondary Outcome: Daily Stool Frequency
Description: Mean change in reported daily stool frequency Analyses of change in daily stool frequency will only include participants with IBS-C and IBS-D. IBS-C and IBS-D subtypes will be analyzed independently.
Time Frame: as for outcome 1
Population: A total of 115 participants treated with GDH are included in the analysis population: 59 patients had IBS-C and 56 patients had IBS-D. A total of 116 patients treated with MR are included: 59 patients had IBS-C and 57 patients had IBS-D. These numbers are smaller than the total size of the IBS-C and IBS-D populations because not all patients completed the daily diaries for weeks 13 through 16.
Measure: Mean (Standard Deviation); unit: number of bowel movements per day
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 115 | 116
number of bowel movements per day
  IBS-C subgroup of participants: number analyzed (Participants) | 59 | 59
  IBS-C subgroup of participants | -0.074 (0.8964) | 0.151 (0.4531)
  IBS-D subgroup of participants: number analyzed (Participants) | 56 | 57
  IBS-D subgroup of participants | -0.325 (0.6915) | -0.455 (1.2904)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The analysis is based on the mixed model repeated measures (MMRM) analysis of variance model for IBS-C participants: parameter = treatment + timepoint + treatment*timepoint + gender + subject error + random Means are the mean daily number of bowel movements for a 24-hour period; Test type: Superiority; p = 0.6793, Mixed Models Analysis; Mean Difference (Final Values) = 0.080, 95% CI 2-sided [-0.301 to 0.460]
Statistical Analysis 2: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The analysis is based on the mixed model repeated measures (MMRM) analysis of variance model for IBS-D participants: parameter = treatment + timepoint + treatment*timepoint + gender + subject error + random Means are the mean daily number of bowel movements for a 24-hour period; Test type: Superiority; p = 0.9468, Mixed Models Analysis; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [-4.904 to 5.249]

6. Secondary Outcome: Health-related Quality of Life Using the IBS Quality of Life (QOL) Instrument
Description: The IBS QOL is a 34 item IBS-specific, validated instrument. The 34 items are summed for a total score and then transformed to 0-100 scale with higher scores indicating better IBS specific quality of life. IBS QOL scores will be compared pre- and post-treatment and the mean difference compared by treatment.
Time Frame: Baseline (Week -4) to 4-weeks post-treatment (Week 16)
Population: Participants that completed the IBS-QoL at Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 165 | 166
score on a scale | 8.075 (19.2567) | 5.816 (23.0150)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The analysis is based on the mixed model repeated measures (MMRM) analysis of variance model: parameter = treatment + timepoint + treatment*timepoint + gender + subject error + random The unstructured covariance matrix was used to model the within-participant correlation. The model-based least square (LS) means and LS mean differences (GDH minus comparator) and associated 95% CIs for each week and overall were estimated; Test type: Superiority; p = 0.5015, Mixed Models Analysis; Median Difference (Final Values) = -1.602, 95% CI 2-sided [-6.282 to 3.077]

7. Secondary Outcome: Percent Overall Work Impairment Due to IBS Based on the Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: Productivity and absenteeism will be evaluated using the patient reported Work Productivity and Activity Impairment (WPAI) General Health score. The WPAI (Reilly 1993) is a 6-question survey of presenteeism (impairment at work / reduced on-the-job effectiveness) and absenteeism (work time missed).
  The WPAI-GH consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS).
  Outcomes are expressed as impairment percentages (0-100%) with higher numbers indicating greater impairment and less productivity (worse outcomes).
Time Frame: Baseline (Week -4) to 4-weeks post-treatment (Week 16)
Population: Participants who completed the WPAI at Week 16 and who were currently employed (working for pay).
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 90 | 87
percentage of impairment | -18.1 (27.59) | -14.4 (25.22)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; "Percent Overall Work Impairment Due to IBS" defined as the percent time missed by not showing up for work, plus the percent time missed while working, and calculated as: Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)]; Test type: Superiority; p = 0.2117, Mixed Models Analysis; Mean Difference (Final Values) = 4.586, 95% CI 2-sided [-2.619 to 11.790]

8. Secondary Outcome: Percent Overall Activity Impairment Due to IBS Based on the Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: Productivity and absenteeism will be evaluated using the patient reported Work Productivity and Activity Impairment (WPAI) General Health score. The WPAI (Reilly 1993) is a 6-question survey of presenteeism (impairment at work / reduced on-the-job effectiveness) and absenteeism (work time missed).
  The WPAI-GH consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS). Overall activity impairment is based on responses to Question 6.
  Outcomes are expressed as impairment percentages (0-100%) with higher numbers indicating greater impairment and less productivity (worse outcomes).
Time Frame: 4-weeks post-treatment (Week 16)
Population: Participants who completed the WPAI at Week 16
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
Number analyzed (Participants) | 164 | 163
percentage of impairment | 42.9 (25.92) | 40.2 (28.06)
Statistical Analysis 1: Comparison: Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD vs MR-1; Muscle Relaxation, Software as a Medical Device - SaMD; The analysis is based on the mixed model repeated measures (MMRM) analysis of variance model: parameter = treatment + timepoint + treatment*timepoint + gender + subject error + random; Test type: Superiority; p = 0.3676, Mixed Models Analysis; Mean Difference (Net) = 2.372, 95% CI 2-sided [-2.793 to 7.537]

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: All adverse events (AEs) will be coded to system organ class (SOC) and preferred terms (PT).
  A treatment-emergent AE (TEAE) is defined as an AE that was not present prior to treatment with the investigational digital device, but appeared following treatment or was present at treatment initiation but worsened during treatment.
  The frequency of TEAEs will be tabulated by preferred term and system organ class. The maximum severity and frequency of TEAEs will be summarized by treatment.
Arm/Group | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/190
Serious Adverse Events (participants affected / at risk) | 1/188 | 0/190
Other Adverse Events (participants affected / at risk) | 6/188 | 2/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD (N=188) | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD (N=190)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Arnold-Chiari malformation (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regulora; Gut-Directed Hypnotherapy Software as a Medical Device - SaMD (N=188) | MR-1; Muscle Relaxation, Software as a Medical Device - SaMD (N=190)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dydpepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT04133519/Prot_SAP_000.pdf